CLINICAL TRIAL: NCT03689153
Title: A Randomized, Placebo-controlled, Double-blind, Single Ascending Dose Study to Investigate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JNJ-63733657 in Healthy Japanese Subjects
Brief Title: A Study of JNJ-63733657 in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CR108522; 63733657EDI1002 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2025-04-28 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: JNJ-63733657 or Placebo (Experimental): Participants will receive a single intravenous (IV) low dose of JNJ-63733657 or matching placebo.
  Interventions: Drug: JNJ-63733657; Drug: Placebo
- Cohort 2: JNJ-63733657 or Placebo (Experimental): Participants will receive a single IV middle dose of JNJ-63733657 or matching placebo.
  Interventions: Drug: JNJ-63733657; Drug: Placebo
- Cohort 3: JNJ-63733657 or Placebo (Experimental): Participants will receive a single IV high dose of JNJ-63733657 or matching placebo.
  Interventions: Drug: JNJ-63733657; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-63733657 — Single ascending IV low, middle, and high dose of JNJ-63733657 will be administered in sequential cohorts. The progression to the next (higher) dose level is dependent on acceptable safety and tolerability profile of JNJ-63733657 obtained after dose administration of the current dose level. The length of time between dosing days of cohorts will be at least 14 days.
Drug: Placebo — Participants will receive matching placebo intravenously.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of JNJ-63733657 following single ascending intravenous (IV) dose administration in healthy Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI; weight [kilogram {kg}]/height [meter square {m^2}]) between 18 and 35 kilogram per meter square (kg/m^2), inclusive, and a body weight greater than 50 kg but less than 110 kg at screening and Day -1. For participants to be enrolled in the highest dose cohort (Cohort 3), additional weight limitations will apply in order not to exceed the total dose of 5 gram (g) JNJ-63733657; the participant weight in the highest dose cohort will be limited
* Women must not be of childbearing potential

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, coagulation, or urinalysis at screening and Day -1 in the opinion of the investigator
* Clinically significant abnormal physical or neurologic examination (including fundoscopy), vital signs, or 12-lead electrocardiogram (ECG) at screening and Day -1 in the opinion of the investigator
* Positive result on hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus (HCV) antibody (antiHCV) positive, or any other clinically active liver disease at screening (per screening evaluations)
* History of human immunodeficiency virus (HIV) antibody positive, tests positive for HIV or tests positive for syphilis at screening
* Mini-Mental State Examination (MMSE) score less than or equal to (<=) 27 at screening

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Approximately 23 weeks
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of JNJ-63733657 | Up to Day 106
  The Cmax is the maximum observed serum concentration.
Time to Reach Maximum Observed Serum Concentration (Tmax) of JNJ-63733657 | Up to Day 106
  The Tmax is defined as actual sampling time to reach maximum observed serum concentration.
Area Under the Serum Concentration-Time Curve from Time Zero to Time to 56 Days (AUC [0-56days]) | 0 hours (Day 1) up to 56 days
  The AUC (0-56days) is the area under the serum concentration versus time curve from time 0 to time to 56 days after the start of infusion.
Area Under the Serum Concentration-Time Curve from Time Zero to the Time Corresponding to Last Quantifiable Serum Concentration (AUC [0-last]) | Up to Day 106
  The AUC (0-last) is the area under the serum concentration-time curve from time zero time to the time corresponding to the last quantifiable serum concentration.
Area Under the Serum Concentration-Time Curve from Time Zero to Infinite Time (AUC [0-infinity]) | Up to Day 106
  The AUC (0-infinity) is the area under the serum concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z); wherein AUC(0-last) is area under the serum concentration-time curve from time zero to last quantifiable time, C(last) is the last observed measurable serum concentration, and lambda(z) is elimination rate constant.
Elimination Rate Constant (Lambda[z]) of JNJ-63733657 in Serum | Up to Day 106
  Lambda(z) is first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Apparent Elimination Half-Life (t1/2) of JNJ-63733657 in Serum | Up to Day 106
  The elimination half-life (t1/2) is the time measured for the serum concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Total Systemic Clearance (CL) of JNJ-63733657 in Serum | Up to Day 106
  Systemic clearance is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by the serum area under the plasma concentration-time curve from time zero to infinite time (AUC[0-infinity]).
Volume of Distribution (Vz) of JNJ-63733657 in Serum | Up to Day 106
  The Vz is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
JNJ-63733657 Concentration in Cerebrospinal Fluid (CSF) | Up to Day 92
  CSF concentration assessments will be done for JNJ-63733657.
Number of Participants with Anti-JNJ-63733657 Antibodies | Up to Day 106
  Number of participants with anti-JNJ-63733657 antibodies will be determined in serum samples.
Percentage Change from Baseline in Total, Free, and Bound tau Biomarker Fragments in CSF | Up to Day 92
  Percentage change from baseline in total, free, and bound tau (phosphorylation site) biomarker fragments in CSF will be evaluated to assess the effect of JNJ-63733657.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Souseikai Fukuoka Mirai Hospital, Fukuoka, Japan